CLINICAL TRIAL: NCT05798793
Title: A Multi-Center, Randomized Phase III Study of Neoadjuvant Anti-PD-1 Immunotherapy Plus TP Chemotherapy Versus TP Chemotherapy or Up-Front Surgery in Resectable Locally Advanced Oral Squamous Cell Carcinoma
Brief Title: Neoadjuvant Anti-PD-1 Immunotherapy With Chemotherapy in Resectable Locally Advanced Oral Squamous Cell Carcinoma
Acronym: NEOPCOSCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital of Stomatology, Wuhan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Gang Chen, Chief physician, Professor, Hospital of Stomatology, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WuhanHStomatology
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Neoadjuvant; Oral squamous cell carcinoma; Anti-PD-1 immunotherapy; Camrelizumab; TP chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgery followed by postoperative RT (No Intervention): The participants will take a radical surgery followed by radiotherapy or chemoradiotherapy if necessary.
- Neoadjuvant TP chemotherapy (Experimental): The participants will receive 2 courses of TP chemotherapy. Then the participants will take a radical surgery followed by radiotherapy or chemoradiotherapy if necessary.
  Interventions: Drug: TP
- Neoadjuvant anti-PD-1 immunotherapy plus TP chemotherapy (Experimental): The participants will receive 3 doses of PD-1 blockade and 2 courses of TP chemotherapy. Then the participants will take a radical surgery followed by radiotherapy or chemoradiotherapy if necessary.
  Interventions: Drug: Camrelizumab plus TP

INTERVENTIONS:
Drug: Camrelizumab plus TP — The participants will receive camrelizumab (200 mg) through intravenous infusion each 2-week cycle, and docetaxel (T) 75 mg/m2, cisplatin (P) 75 mg/m2 through intravenous infusion each 3-week cycle for 2 cycles.
  Other Names: SHR-1210 plus Docetaxel, Cisplatin
  Arms: Neoadjuvant anti-PD-1 immunotherapy plus TP chemotherapy
Drug: TP — The participants will receive docetaxel (T) 75 mg/m2, cisplatin (P) 75 mg/m2 through intravenous infusion each 3-week cycle for 2 cycles.
  Other Names: Docetaxel, Cisplatin
  Arms: Neoadjuvant TP chemotherapy

SUMMARY:
The purpose of this study is to investigate the survival benefit of neoadjuvant anti-PD-1 immunotherapy plus TP chemotherapy compared with TP chemotherapy or up-front surgery in resectable locally advanced oral squamous cell carcinoma.

DETAILED DESCRIPTION:
On the basis of preliminary study, this study is to further verify the efficacy and safety of neoadjuvant anti-PD-1 immunotherapy plus chemotherapy. The further purpose of this study is to investigate the survival benefit of neoadjuvant anti-PD-1 immunotherapy plus TP chemotherapy compared with TP chemotherapy or up-front surgery in resectable locally advanced oral squamous cell carcinoma. And on this basis, the investigators will explore the changes of the profiles and functions of immune cells within tumors, lymph nodes and peripheral blood after the experimental interventions, as well as their correlation with the patients' response and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented oral squamous cell carcinoma (biopsy required).
2. Local advanced oral squamous cell carcinoma (clinical stage T1-2N1-2M0, T3-4aN0-2M0) with resection option for potential cure, as assessed by a faculty surgeon at Hospital of Stomatology, Wuhan University.
3. Distant metastasis is excluded by chest CT and emission computed tomograph.
4. Adequate organ function as follows: 1) Leukocyte count ≥ 2,000/mm3; 2) Absolute neutrophil count ≥ 1,000/mm3; 3) Platelet count ≥ 100,000/mm3; 4) Hemoglobin ≥ 90 g/L; 5) Serum albumin ≥30 g/L; 6) Total bilirubin ≤ 1.5 × upper limit of normal (ULN); 7) AST (SGOT) and ALT (SGPT) < 2.5 × ULN; 8) ALP ≤ 2.5 × ULN; 9) Prothrombin time-international normalized ratio ≤ 1.5; 10) Serum creatinine ≤ 1.5 × ULN; 11) INR/PT≤ 1.5; 12) TSH ≤ ULN.
5. ECOG performance status 0-1.
6. Female patient tested HCG negative in serum or urine within 7 days prior to the start of investigational product. Both patient and partner must agree to use contraception prior to study entry and for the duration of study participation and for up to 120 days after the last dose of PD-1 blockade.
7. Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form.

Exclusion Criteria:

1. History of ≥ 3 grade immune related adverse events (irAEs) or have not recovered to ≤ 1 grade irAEs from previous treatment.
2. History of other treatments for cancer, including surgery, chemotherapy, radiotherapy or molecular targeted therapy within past 5 years.
3. Previous therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 or any other antibody targeting T cell co-regulatory pathways.
4. Active autoimmune disease or history of refractory autoimmune disease.
5. Active systemic infection requiring therapy.
6. Patients who are receiving psychotropic drug or alcohol/drug abuse.
7. Subjects with concurrent other active malignancies.
8. HIV or untreated active HBV or HCV infections, or vaccinated (HBV, flu, varicella, etc) within 4 weeks before recruitment.
9. Uncontrollable systemic diseases, including diabetes, hypertension, etc.
10. History of stroke or transient ischemic attack within past 6 months.
11. Distant metastases or inability to resect after physician evaluation.
12. Serious cardiovascular, respiratory, immune system critical disease or other conditions that the researchers thought might increase the subjects' risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) Rate on Each Treatment Arm. | 24 months.
  EFS is the time from the date of randomization to the date of first record of disease progression as defined by RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) on Each Treatment Arm. | 24 months.
  OS is the time from randomization to death due to any cause.
Radiographic Response. | 8 weeks.
  Clinical response of tumors and lymph nodes to neoadjuvant PD-1 blockade alone or neoadjuvant PD-1 blockade plus TPF induction chemotherapy, as evaluated by radiographic examinations and defined by RECIST 1.1.
  Clinical response of tumors and lymph nodes to neoadjuvant PD-1 blockade alone or neoadjuvant PD-1 blockade plus TPF induction chemotherapy, as evaluated by radiographic examinations and defined by RECIST 1.1.
Pathologic Response. | 8 weeks.
  Pathologic response of resected tumors and lymph nodes to neoadjuvant PD-1 blockade alone or neoadjuvant PD-1 blockade plus TPF induction chemotherapy. Pathologic response is defined as sum of pathologic complete response and major pathologic response. Pathologic complete response is defined as the absence of viable residual tumor in resected specimen. The rate of major pathologic response, defined as <10% residual viable tumor cells in the resected specimen.
Adverse Events (AEs). | 24 months.
  Number of participants experiencing any sign, symptom, disease, or worsening of preexisting conditions temporally associated with the experimental interventions or irrespective of the experimental interventions.

OTHER OUTCOMES:
Changes in the Level of Circualting Exosomal PD-L1. | 24 months.
  The level of circulating exosomal PD-L1 at serial time points pre- and on-treatment, as detected by enzyme-linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, M.D., Principal Investigator — Hospital of Stomatology, Wuhan University
Locations (3):
- China (3):
  - Peking university Shenzhen hospital, Shenzhen, Guangdong
  - Hospital of Stomatology, Wuhan University, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No